CLINICAL TRIAL: NCT07313293
Title: Impact of Foot Reflexology on Nausea After Obesity Surgery
Acronym: IRANNO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD25_0097
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sleeve Gastrectomy
Keywords: foot reflexology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care alone (No Intervention)
- Conventional care + foot reflexology (Experimental)
  Interventions: Other: Foot reflexology

INTERVENTIONS:
Other: Foot reflexology — Foot reflexology sessions to:
  * Prepare the body and mind for surgery
  * Promote physical and nervous relaxation
  * Relieve post-operative nausea and vomiting
  Arms: Conventional care + foot reflexology

SUMMARY:
Obesity is a major public health issue. The Obépi epidemiological survey, the results of which were published in 2020, shows a steady increase in obesity among the French population.

Currently, more than 23 million French people are overweight or obese, and more than 8 million French people are obese. The most effective treatment currently available is surgery. These procedures are governed by specific recommendations. Between 50,000 and 60,000 procedures are performed in France each year. Three procedures are authorised: gastric banding, sleeve gastrectomy and gastric bypass.

Hallyday & al report 65% of patients experiencing nausea/vomiting after bariatric surgery. In 2019, Suh & al showed that nausea and vomiting were more common after sleeve gastrectomy and that they were responsible for an increase in the length of hospitalisation. These episodes of nausea and vomiting occur within 48 hours after sleeve gastrectomy and can cause difficulties in resuming eating. One of the factors contributing to the occurrence of nausea and vomiting was the use of opioids.

The benefits of foot reflexology were reported in 2023 by Dr Carrazé in rectal surgery. His doctoral thesis in medicine showed that foot reflexology sessions on days 1, 2 and 3 following rectal surgery reduced post-operative ileus and post-operative pain. The reduction in post-operative ileus led to a decrease in episodes of nausea and vomiting.

In 2021, Murat-Ringot & al demonstrated the beneficial effect of foot reflexology on nausea and vomiting during chemotherapy sessions, in addition to the anti-emetic treatments used for prevention. Anderson & al. in 2021 also demonstrated a beneficial effect on pain in cancer patients, with no effect on nausea.

The principle of foot reflexology is based on the fact that each organ, gland or part of the body corresponds to a reflex zone on the foot, hand, ears or face. Stimulation of the reflex zones is thought to activate the autonomic nervous system. Currently, there is very little scientific evidence on how this practice works and what its effects are. Despite various scientific publications on the results of foot reflexology, scientific evidence of its effectiveness remains weak. Only one prospective randomised trial has been found in the literature (Dalal & al.) on the quality of life of patients with epilepsy.

Despite the lack of high-quality studies, it appears that foot reflexology could benefit patients by reducing nausea and vomiting. To date, no studies have evaluated its effectiveness in the post-operative period, particularly after bariatric surgery.

The aim of our randomised trial is to evaluate the impact of foot reflexology on nausea and vomiting after sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient scheduled to undergo sleeve gastrectomy
* Patient capable of understanding the protocol and having given their informed verbal consent to participate in the study
* Patient affiliated with the social security system or entitled to benefits

Exclusion Criteria:

* Patients receiving long-term morphine and opioid treatment
* Patients with phlebitis, a wound under the foot, or recent foot trauma (cast immobilisation, splint, etc.)
* Patients under guardianship, curatorship, or deprived of their liberty
* Patients who are pregnant, breastfeeding, or refusing contraception
* Patients participating in another clinical research protocol that has an impact on the objective of the study
* Patients under an activated future protection mandate
* Patients under family authorisation
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2028-02-03 (Estimated); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing significant nausea and/or vomiting (with a score ≥ 3 on a numerical scale of 0 to 10) within 24 hours post-operatively | 24 hours post-operatively
  A score of ≥ 3 corresponds to the introduction of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Principal Investigator — Centre Hospitalier Departemental Vendee
Locations (1):
- Centre Hospitalier Départemental Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalal K, Devarajan E, Pandey RM, Subbiah V, Tripathi M. Role of reflexology and antiepileptic drugs in managing intractable epilepsy--a randomized controlled trial. Forsch Komplementmed. 2013;20(2):104-11. doi: 10.1159/000350047. Epub 2013 Apr 15. PMID 23636029
- [Background] Anderson KD, Downey M. Foot Reflexology: An Intervention for Pain and Nausea Among Inpatients With Cancer. Clin J Oncol Nurs. 2021 Oct 1;25(5):539-545. doi: 10.1188/21.CJON.539-545. PMID 34533507
- [Background] Murat-Ringot A, Souquet PJ, Subtil F, Boutitie F, Preau M, Piriou V. The Effect of Foot Reflexology on Chemotherapy-Induced Nausea and Vomiting in Patients With Digestive or Lung Cancer: Randomized Controlled Trial. JMIR Cancer. 2021 Nov 5;7(4):e25648. doi: 10.2196/25648. PMID 34738909
- [Background] Suh S, Helm M, Kindel TL, Goldblatt MI, Gould JC, Higgins RM. The impact of nausea on post-operative outcomes in bariatric surgery patients. Surg Endosc. 2020 Jul;34(7):3085-3091. doi: 10.1007/s00464-019-07058-5. Epub 2019 Aug 6. PMID 31388805
- [Background] Halliday TA, Sundqvist J, Hultin M, Wallden J. Post-operative nausea and vomiting in bariatric surgery patients: an observational study. Acta Anaesthesiol Scand. 2017 May;61(5):471-479. doi: 10.1111/aas.12884. PMID 28374473